CLINICAL TRIAL: NCT04213560
Title: The Effects of Weighted Waist-Hooping on Balance, Proprioception, and Body Awareness
Brief Title: The Effects of Weighted Waist-Hooping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Sage Colleges (Other)
Responsible Party: Principal Investigator, Brittney Muir, Assistant Professor, The Sage Colleges
Organization: VA Puget Sound Health Care System (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 545-2016-2017
Record Dates: First submitted 2019-12-18; First posted 2019-12-30 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Weighted waist-hooping; Balance; Proprioception; Neurocom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted waist-hooping (Experimental): Participants weighted waist-hooping on their own for ten minutes a day, four days a week, for six weeks resulting in a total of 40 minutes of weighted waist-hooping each week. Participants weighted waist-hooped with a three-pound weighted hula hoop at the waist for ten minutes. Half time hooping to the left and the other half hooping to the right. If discomfort while hooping occurred participants were instructed to take breaks, change directions more frequently, or where thicker clothing to lessen the impact of the hoop around their waists. The investigators would check in on the participants weekly to provide feedback on technique and answer all questions throughout the six-week intervention.
  Interventions: Device: weighted waist-hooping
- Control (No Intervention): No Intervention

INTERVENTIONS:
Device: weighted waist-hooping — weighted waist-hooping
  Arms: Weighted waist-hooping

SUMMARY:
Purposes: 1) To determine the effects of weighted waist-hooping on balance in healthy individuals and 2) to observe whether these effects are attributed to neuromuscular conditioning or core strength gains.

Methods: 27 females (ages 20-45) were included, 15 in the intervention group, and 12 in the control. The intervention consisted of six weeks of weighted waist-hooping four times a week for 10 minutes each session. Balance was assessed pre and post intervention using the BESS, SEBT, and Neurocom SOT. Core strength was assessed using hold duration of a bilateral and unilateral plank.

ELIGIBILITY:
Inclusion Criteria:

* healthy women age 18-45.

Exclusion Criteria:

* pregnancy and vertigo

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Balance Error Scoring System (BESS) | baseline
  Participants were instructed to maintain each of the 6 positions for as long as possible and to continue to try until the 20 seconds were complete even if balance was lost, which was counted as an error along with the specific error criteria for this assessment. Total number of errors were recorded for each position according and the summated to provide a total error score. A higher score indicates greater occurrence of error and thus poorer balance.
Balance Error Scoring System (BESS) | 6 - weeks
  Participants were instructed to maintain each of the 6 positions for as long as possible and to continue to try until the 20 seconds were complete even if balance was lost, which was counted as an error along with the specific error criteria for this assessment. Total number of errors were recorded for each position according and the summated to provide a total error score. A higher score indicates greater occurrence of error and thus poorer balance.
Star Excursion Balance Test (SEBT) | baseline
  SEBT was conducted for both the right and left leg reaching. Position on the start was used to indicate where to reach. Reaching across the body with the right foot to the left side and reaching across the body with the left foot to the right side were both defined as a medial reach for the purpose of this study.
Star Excursion Balance Test (SEBT) | 6 - weeks
  SEBT was conducted for both the right and left leg reaching. Position on the start was used to indicate where to reach. Reaching across the body with the right foot to the left side and reaching across the body with the left foot to the right side were both defined as a medial reach for the purpose of this study.
equilibrium scores (EQ scores) of the Sensory Organization Test (SOT) on the NeuroCom | baseline
  The SOT parses out contributions and functionality of the visual, somatosensory, and vestibular systems provide information regarding the effects of each system on postural control.8 The EQ score is a composite score calculated by the NeuroCom by weighting each of the 6 conditions of typical and altered stimuli. A score closer to 100 indicates less postural sway and a score closer to 0 indicates more postural sway and increased likelihood of fall.8 An increase in EQ score indicates an improvement in postural control and potentially sensory selection since the purpose of the SOT is to determine if patients are able to appropriately reweight their senses in response to the six different conditions in an effort to maintain postural control.
equilibrium scores (EQ scores) of the Sensory Organization Test (SOT) on the NeuroCom | 6 - weeks
  The SOT parses out contributions and functionality of the visual, somatosensory, and vestibular systems provide information regarding the effects of each system on postural control.8 The EQ score is a composite score calculated by the NeuroCom by weighting each of the 6 conditions of typical and altered stimuli. A score closer to 100 indicates less postural sway and a score closer to 0 indicates more postural sway and increased likelihood of fall.8 An increase in EQ score indicates an improvement in postural control and potentially sensory selection since the purpose of the SOT is to determine if patients are able to appropriately reweight their senses in response to the six different conditions in an effort to maintain postural control.
Core Strength position 1 | baseline
  hold a standard bilateral plank position to assess core strength. The duration of time the participant was able to hold each position was recorded. If the participant was unable to attain proper form or unable to complete the task the duration of hold was recorded as 0 seconds. These assessments were conducted before and after the weighted waist-hooping intervention.
Core Strength position 1 | 6 - weeks
  hold a standard bilateral plank position to assess core strength. The duration of time the participant was able to hold each position was recorded. If the participant was unable to attain proper form or unable to complete the task the duration of hold was recorded as 0 seconds. These assessments were conducted before and after the weighted waist-hooping intervention.
Core Strength position 2 | baseline
  hold a unilateral plank with the dominant leg raised position to assess core strength. The duration of time the participant was able to hold the position was recorded. If the participant was unable to attain proper form or unable to complete the task the duration of hold was recorded as 0 seconds. These assessments were conducted before and after the weighted waist-hooping intervention.
Core Strength position 2 | 6 - weeks
  hold a unilateral plank with the dominant leg raised position to assess core strength. The duration of time the participant was able to hold the position was recorded. If the participant was unable to attain proper form or unable to complete the task the duration of hold was recorded as 0 seconds. These assessments were conducted before and after the weighted waist-hooping intervention.

IPD SHARING:
Plan to Share IPD: No